CLINICAL TRIAL: NCT05817877
Title: Investigation of the Relationship of Smartphone Use Time With Neck Endurance, Head Posture, Lateral Grip Strength, Hand Grip Strength and Postural Control Parameters in Young Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Zeynep SAG, physiotherapist, Dokuz Eylul University
Other Study IDs: 2023/03-14
Record Dates: First submitted 2023-03-23; First posted 2023-04-18 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Cell Phone Use
Keywords: CoP; Balance; forehead posture
MeSH Terms: conditions — Cell Phone Use

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- over 5 hours: people with an average daily phone use of more than 5 hours.
  Interventions: Other: phone use
- under 5 hours: People with an average daily phone use of less than 5 hours.
  Interventions: Other: phone use

INTERVENTIONS:
Other: phone use — There is no intervention.

SUMMARY:
In the planned study, young adults between the ages of 18-35 with different phone usage durations will be evaluated. The aim of the study is to investigate whether the average daily phone usage time has a direct relationship with neck muscle endurance, rough grip strength, lateral grip strength and head posture, and whether there is an indirect relationship with postural control. People who have phones with IOS 12 or Android 9 and above will be invited to the study. By looking at the screen time tracking feature in these versions, the daily phone usage hour for the last week will be calculated and the participants will be divided into two groups as the daily phone usage average of 5, and below and 5 hours. In the planned study, neck endurance will be tested on flexor and extensor muscle groups in accordance with the literature. The lateral flexion and anterior tilt angles will be calculated with two photographs taken from the anterior and lateral sides of the head posture of the person's shoulder, and the hand grip strength will be measured with a Jamar hand dynamometer and the lateral grip strength will be measured with a pinchmeter. Postural control evaluation will be measured by means of center of pressure-CoP parameters measured with TekScan brand pressure platform. The study is planned to be carried out in the Movement Analysis Laboratory of the Faculty of Physical Therapy and Rehabilitation of Dokuz Eylul University. Participants will be selected from healthy adults between the ages of 18-35 who volunteered to participate in the study among the students of the Faculty of Physical Therapy and Rehabilitation, their relatives and the relatives of the researcher. The study is planned to be completed within 6 months following ethical approval.

ELIGIBILITY:
Inclusion Criteria:

* Using a phone with IOS 12 or android 9 and above for at least one week

Exclusion Criteria:

* Presence of orthopedic surgery in the last 6 months
* Those who have a disease or take medication that will prevent neuromuscular system and postural control measurements
* have neck pain

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy young adults
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2024-03-14 (Estimated)

PRIMARY OUTCOMES:
postural control parameters | up to 8 weeks
  Postural control can be quantitatively assessed by examining the behavior of the statically or dynamically in the lower pressure center (CoP).

SECONDARY OUTCOMES:
hand grip strength | up to 8 weeks
  hand grip is the numerical output of the brute grip strength of the hand
lateral grip strength | up to 8 weeks
  The lateral grip is a numerical measurement of the maximum strength of the thumb abductor muscles, which we do not use especially during texting.
neck muscle endurance | up to 8 weeks
  neck muscle endurance is the numerical data of the endurance of the neck flexor and extensor muscles

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylül Univercity, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes